CLINICAL TRIAL: NCT00846612
Title: Phase II and Pharmacokinetic Study of Avastin and Doxil in the Treatment of Platinum-resistant or Refractory Ovarian Cancer
Brief Title: Pharmacokinetic Study of Avastin and Doxil in Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Genentech, Inc. (Industry); University of New Mexico Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-948; Genentech AVF3910s (Other: Genentech)
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Cancer
Keywords: refractory; avastin; doxil; relapsed; ovarian cancer; platinum-resistant
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — liposomal doxorubicin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Avastin-Doxil (Experimental)
  Interventions: Drug: Doxil; Drug: Bevacizumab (Avastin)

INTERVENTIONS:
Drug: Doxil — 1 cycle: 3 weeks; 30 mg/m^2, IV, every cycle
  Other Names: pegylated doxorubicin liposome
Drug: Bevacizumab (Avastin) — 1 cycle: every 3 weeks; 15 mg/kg, IV, beginning on cycle 2 and every cycle 20-24 hours following Doxil administration
  Other Names: Avastin

SUMMARY:
This study is to study pharmacokinetics of Doxil using Doxil and Avastin on ovarian cancer patients who are resistant to or have relapsed from platinum-based therapy.

DETAILED DESCRIPTION:
This study registration at clinicaltrials.gov is divided into 2 records. This record (NCT00846612) is for pharmacokinetics of Doxil. Another record (NCT00945139) describes the efficacy and safety of the combination treatment.

Treatment upon diagnosis of epithelial ovarian cancer (EOC) consists of surgery to achieve maximal tumor debulking followed by platinum-based chemotherapy (carboplatin + paclitaxel). Recently, optimally (e.g., < 1 cm residual disease) debulked patients appear to benefit from regimens that include intraperitoneal administration of cisplatin. While complete response (CR) is frequently achieved, by two years 50% of the patients show signs of recurrence.

When EOC presenting at an advanced stage recurs, even after a CR had been achieved, it can no longer be totally eradicated. Nevertheless, a number of drugs lead to objective responses, patients benefit with a prolongation of survival. Anti-tumor activity of Doxil against ovarian cancer was noted in a phase I study, and this was followed by a phase II study that demonstrated activity in platinum and paclitaxel refractory disease. In the expanded phase II experience at the University of Southern California, responses to Doxil occurred preferably in disease that was not bulky and after fewer prior treatments. Typically, several cycles were required for maximum response, and some patients had prolonged stable disease. Subsequently, the study of Gordon et al established the preferred role of this drug formulation in the 2nd line-setting. It is logical, therefore, to build on this agent in trying to improve the outcome of patients with recurrent ovarian cancer, and in particular, to consider a combination with Avastin, since Avastin has shown agent activity in retrospective data and recent studies in EOC.

A combination of Doxil with Avastin has several aspects of interest to ovarian cancer treatment: 1) independent single-agent activity, 2) enhanced localization of Doxil is possible via increased half-life (if liposomal egress is diminished) and decreased tumoral interstitial pressure, 3) improved Doxil distribution, and 4) likely favorable toxicity profile since Doxil's only common problematic toxicity is to the skin (palmar-plantar erythrodysesthesia or PPE). Pharmacokinetic issues will be addressed in selected patients, by comparing cycle 1 (without Avastin) with cycle 2 (with Avastin).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be platinum resistant
* No prior anthracycline use
* PS ≤ 2
* Lab values within certain limits (ANC > 1000, platelets > 100,000; ALT, AST 2x ULN, creatinine < 2.0);
* No more than 3 prior chemotherapy regimens, only 2 of which can have included platinum-containing regimens.
* Use of effective means of contraception in subjects of child-bearing potential

Exclusion Criteria:

* Disease-Specific Exclusions:

  * Evidence of complete or partial bowel obstruction
  * Need for IV hydration or TPN
  * > 2 prior abdominal surgeries
  * History of gastrointestinal perforation
  * Gastrointestinal perforation due to any other cause within the last 6 months
* General Medical Exclusions:

  * Inability to comply with study and/or follow-up procedures
  * Life expectancy of less than 12 weeks
  * Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin cancer study
* Avastin-Specific Exclusions:

  * Inadequately controlled hypertension (defined as systolic blood pressure greater than 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
  * Any prior history of hypertensive crisis or hypertensive encephalopathy
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E of the protocol)
  * History of myocardial infarction or unstable angina within 6 months prior to study enrollment
  * History of stroke or transient ischemic attack within 6 months prior to study enrollment
  * Known CNS disease
  * Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
  * Symptomatic peripheral vascular disease
  * Evidence of bleeding diathesis or coagulopathy
  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
  * Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
  * History of abdominal fistula, or intra-abdominal abscess within 6 months prior to study enrollment
  * Serious, non-healing wound, ulcer, or bone fracture
  * Proteinuria at screening as demonstrated by either

    * Urine protein:creatinine (UPC) ratio no less than 1.0 at screening OR
    * Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
  * Known hypersensitivity to any component of Avastin
  * Pregnant (positive pregnancy test) or lactating. No effective means of contraception (men and women) in subjects of child-bearing potential

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
change in peak plasma concentration of Doxil without and with Avastin | 1 hour, 1, 4, 7, 10, 14, and 21 days post-dose in cycle 1 and cycle 2
  In cycle 1, patients were treated only with Doxil; in cycle 2, patients were treated with Doxil and Avastin.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Muggia, MD, Principal Investigator — NYU Langone Health
Locations (4):
- United States (4):
  - Univ. of New Mexico cancer research and treatment center, Albuquerque, New Mexico
  - Bellevue Hospital, New York, New York
  - NYU Cancer Center, New York, New York
  - NYU medical center (Tisch Hospital), New York, New York